CLINICAL TRIAL: NCT07008781
Title: A Youth-led Intervention to Reduce Healthcare Disparities in Cancer Screening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sara Heinert, PhD, MPH, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2025000586
Record Dates: First submitted 2025-05-05; First posted 2025-06-06 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: cancer screening; adolescents; high school; community-based research; community health; Hispanic/Latino community
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth-led cancer screening intervention (Experimental): High school students will be trained as health advocates and then facilitate discussions about cancer screening recommendations and risk factors with adults in their community. High school students (15-18 years old) from the local community will be recruited for this study, and each student will recruit adults that they live with or are part of their community (i.e. parent) who are eligible for cancer screening. The adult plus youth dyads will all undergo the same youth-led intervention in which the youth will utilize motivational interviewing to discuss cancer screening recommendations and risk factors with their adults and help their adults enroll in cancer screening through ScreenNJ, a community organization that aims to increase cancer screening in New Jersey, reduce cancer mortality rates, and reduce disparities.
  Interventions: Behavioral: Youth-led cancer screening intervention

INTERVENTIONS:
Behavioral: Youth-led cancer screening intervention — High school students will be trained as health advocates and then facilitate discussions about cancer screening recommendations and risk factors with adults in their community. High school students (15-18 years old) from the local community will be recruited for this study, and each student will recruit adults that they live with or are part of their community (i.e. parent) who are eligible for cancer screening. The adult plus youth dyads will all undergo the same youth-led intervention in which the youth will utilize motivational interviewing to discuss cancer screening recommendations and risk factors with their adults and help their adults enroll in cancer screening through ScreenNJ, a community organization that aims to increase cancer screening in New Jersey, reduce cancer mortality rates, and reduce disparities.

SUMMARY:
This study engages youth as health advocates to increase cancer screening in their community. The study will evaluate the effectiveness of a youth-led intervention on cancer screening awareness in adults who are overdue for cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Student at New Brunswick Health Sciences Technology High School (15-18 years) and their adult family members (18+ years old) who are NJ residents.
* Adults must be eligible for at least one cancer screening other than skin (see below).
* Participants must be fluent in either English or Spanish and the youth must speak the same language as the adult.

Breast: 40-74 year old women Cervical: 21-65 year old women with a cervix (have not had a hysterectomy) Colorectal: 45-75 year olds Prostate: 50 to 69 year old men (start at 45 for black males) Lung: 50 to 80 year olds who currently smoke or quit within the past 15 years

Overall:

21-75 year old women 45-75 year old men 76-80 year olds who currently smoke or quit within the past 15 years

Exclusion Criteria:

* Students less than 15 years old.
* Adults not eligible for a cancer screening of interest.
* Unable to speak fluent English or Spanish.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Rate of Cancer Screening | 2 weeks post-intervention
  % of adults who schedule or conduct cancer screening 2 weeks post-intervention

SECONDARY OUTCOMES:
Change in Cancer Screening Knowledge- Adult | Baseline and 3 days later
  Change in Pre-/post-cancer screening knowledge in the adult using a 7-item assessment that the study team created. Higher scores indicate more knowledge.
Change in Cancer Screening Knowledge- Youth | Baseline and after intervention ends
  Change in Pre-/post-cancer screening knowledge in the youth using a 7-item assessment that the study team created. Higher scores indicate more knowledge.
Change in Youth Self-Efficacy | Baseline and after intervention ends
  Change in Pre-/post youth self-efficacy using a 10-item assessment that the study team created and includes some questions adapted from Patient Activation Measure (PAM-10). Higher scores indicate more self-efficacy.
Change in Adult Activation | Baseline and 3 days later
  Change in Pre-/post adult activation using a 5-item assessment adapted from Patient Activation Measure (PAM-10). Higher scores indicate more activation.
Proportion of adults who are overdue for each cancer type | Baseline
  Proportion of adults who are overdue for each cancer type

CONTACTS AND LOCATIONS:
Locations (1):
- New Brunswick Health Sciences Technology High School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No